CLINICAL TRIAL: NCT02010424
Title: Multicentric Clinical Trial to Improve Blastocyst Utilisation Rate (in Relation to 2 PN Embryos) by Group Culture of Human Embryos in WOW Dishes.
Brief Title: Evaluation of Group Culture in WOW Dishes of Human Embryos in Order to Optimize the Single Embryo Transfer (SET) Strategy.
Acronym: WOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/819
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Fertility
Keywords: reduced fertility
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual culture (Experimental): standard IVF protocol: half of the fertilized oocytes of the patient will be cultured individually in drops of 25 µl Cook cleavage medium till day 3 after fertilization and subsequently in drops of 25 µl Cook blastocyst medium till day 5 after fertilization
  Interventions: Other: control group
- WOW (Experimental): Half of the fertilized oocytes of the patient will be cultured in group in a WOW dish, each in a separate microwell but covered with one drop of 30 µl of Cook cleavage medium till day 3 after fertilization and subsequently all the embryos will be transferred to a new WOW dish (in the exactly the same position) covered with 30 µl of Cook blastocyst medium till day 5 after fertilization
  Interventions: Device: Primo Vision embryo culture dish (CE labeled, Vitrolife)

INTERVENTIONS:
Other: control group — standard IVF protocol
  Arms: Individual culture
Device: Primo Vision embryo culture dish (CE labeled, Vitrolife)
  Arms: WOW

SUMMARY:
In cattle less than 10% of the embryos develop to the blastocyst stage when embryos are cultured individually, however when bovine embryos are cultured in groups a typical 25-35% of blastocysts can be observed. This tendency, i.e. improved embryo development in group culture, has also been demonstrated in other mammalian species, such as mouse, cat and human. The main reason for this beneficial outcome of group culture has been ascribed to the presence of autocrine factors, which are factors secreted by preimplantation embryos that act upon the embryo itself or the neighboring embryos .

Although group culture systems are common in in vitro production systems for animal embryos, it is rarely done in human settings, where individual follow-up of the embryo during the whole culture period is of utmost importance. Recently a CE-labelled culture device has been designed for human embryos, that allow to combine the benefits of both group culture approaches and individual culture. The WOW dish is commercially available by Primo Vision and consists of 9 small microwells on the bottom of the plate, so that the embryos can be cultivated individually in a microwell, but covered by the same drop of culture medium.

In this clinical randomized trial, 158 patients will be included of which half of the fertilized oocytes will be cultured individually (standard culture system) and half of the fertilized oocytes will be cultured in group in a WOW dish, both during five days of culture. The aim of this study is to increase the number of blastocysts suitable for transfer or cryopreservation by culturing the embryos in WOW dishes.

ELIGIBILITY:
Inclusion Criteria:

* Sperm obtained by ejaculation
* Conventional IVF/ICSI
* At least 10 fertilized oocytes (2 PN)

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Blastocyst utilisation rate | 5 days after fertilization
  number of blastocysts out of fertilized oocytes observed 5 days after fertilization that can be used for the patient (fresh transfer or cryopreservation)

SECONDARY OUTCOMES:
Morphologic evaluation | 5 days after fertilization
  Morphologic evaluation according to the Gardner score (Gardner and Schoolcraft, 1999)
change in embryo development | at day 2, 3 and 4 after fertilization
  morphologic evaluation at day 2, 3 and 4 after fertilization
pregnancy rate | day 15 and week 5 after embryo transfer
  endocrine pregnancy by measuring hCG in blood sample on day 15 after embryo transfer and clinical pregnancy confirmed by ultrasound, 5 weeks after embryo transfer.
life birth rate | 9 months after embryo transfer
  birth of a baby nine months after embryo transfer
change in secretome | day 3 and day 5 after fertilization
  embryo conditioned medium will we collected at day 3 and day 5 after fertilization in eppendorf tubes and kept in -80°C until all samples are collected and they will be analyzed with mass spectrometry to compare the secretome (secreted proteins by the preimplantation embryo).

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Antwerp University Hospital, Centre for Reproductive Medicine, Edegem
  - Ghent University Hospital, Ghent